CLINICAL TRIAL: NCT04188990
Title: Evaluation of the Effectiveness and Cost Effectiveness of an Intervention in Hospitalized Patients With Disease-related Malnutrition
Brief Title: Cost Effectiveness of an Intervention in Hospitalized Patients With Disease-related Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, JOSE M QUINTANA-LOPEZ, MD PhD, Head of Research Unit, Hospital Galdakao-Usansolo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI18/00698
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pancreatitis, Acute; Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases; Pancreatic Cancer; Esophagus Cancer; Gastric Cancer; Colorectal Cancer
Keywords: disease-related malnutrition; effectiveness; cost effectiveness
MeSH Terms: conditions — Pancreatitis; Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: After hospital admission, a nutritional screening in all patients who fulfill the selection criteria of the selected centers will be performed. The first branch includes an intervention in the groups of patients who, after screening, are identified as having disease-related malnutrition (DRM) or at risk of DRM, and a follow-up of the rest of the patients; a second cohort / branch will include patients in whom the intervention, if given, is performed by demand by the medical staff responsible for each patient. The third branch / cohort where usual hospital practice will be provided without any explicit nutritional intervention, except the screening to be carried out in all branches
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm (Active Comparator): The "Intervention arm" includes an intervention in the groups of patients who, after screening, are identified as having disease-related malnutrition (DRM) or at risk of DRM, and a follow-up of the rest of the patients
  Interventions: Dietary Supplement: Nutritional dietary intervention
- By demand arm (Placebo Comparator): The "By demand arm" will include patients in whom the nutritional intervention, if given, is performed by demand by the medical staff responsible for each patient.
  Interventions: Dietary Supplement: By demand
- Usual care arm (Placebo Comparator): In the "Usual care arm" usual hospital practice is followed without any explicit nutritional intervention
  Interventions: Dietary Supplement: Usual current care

INTERVENTIONS:
Dietary Supplement: Nutritional dietary intervention — The intervention will be carried out by the Endocrinology and Nutrition Service of hospital 1, where the type of therapeutic action to be developed will be established (Dietary advice, Oral Nutritional Supplementation (SNO), Enteral Feeding or Parenteral Nutrition). The Total Calorie Balance, calories from feeding or with Oral Nutritional Supplementation (ONS), enteral, parenteral, and protein intake will be recorded. The steps to be taken are the following: A.-In patients with preserved oral intake capacity apply the most appropriate dietary measures in each case. B.-If the oral route is contraindicated, it will be assessed if it is possible to use the gastrointestinal tract and enteral nutrition will begin until the patient recovers the oral intake capacity. C.-If the use of the gastrointestinal tract is not indicated, parenteral nutrition will be assessed until digestive function is restored.
  Arms: Intervention arm
Dietary Supplement: By demand — In the "By demand" arm, it is by clinical judgement of the doctor responsible of each patient that can be demanded a nutritional intervention to the nutrition unit of the center's endocrinology service that will judge the type of intervention. This is their usual care right now
  Arms: By demand arm
Dietary Supplement: Usual current care — In th "Usual care" arm, there is no explicit nutritional intervention performed at this time for those patients and, therefore, their usual regular nutritional care will be provide
  Arms: Usual care arm

SUMMARY:
Objectives: To evaluate the effectiveness, and cost-effectiveness, of three hospitalized patient care strategies in relation to disease-related malnutrition (DRM) hospital admissions based on results such as length of stay of the index admission, and from admission until one year after admission, mortality rate, appearance of complications, changes in weight and nutritional state, changes in their health related quality of life and functional status, readmissions, use of health services resources (primary care, hospital and emergency consultations) and costs. Methodology: Intervention study involving three hospitals with three branches in which, after nutritional screening in all centers, the first branch / hospital includes a intervention strategy for nutritional improvement in patients who after screening are identified as having DRE or at risk of DRE, and follow-up of other patients; a second cohort / hospital will include similar patients in which if there is any nutritional intervention it will be carried out by demand of the medical staff in charge of the patient; and a third branch /hospital in which the usual practice of the center will be followed without any explicit intervention. Subjects of the study: At least 300 patients in each center admitted to the digestive services, due to digestive pathologies, and surgery services due to tumor and digestive system pathologies. In all patients, sociodemographic and clinical data will be collected and of the outcomes described above during admission and until the year of follow-up. Statistical analysis: through appropriate multiple regression models for each outcome variable and with adjustments through propensity scores to compare the three centers based on each outcome parameter. A cost-effectiveness analysis will be carried out through of the incremental cost for each year of quality-adjusted life (QALY) .

DETAILED DESCRIPTION:
Objectives

1. -After a nutritional screening of all patients, evaluate the effectiveness of an intervention in patients admitted to a hospital in relationship to disease-related malnutrition (DRM) by comparing 3 cohorts: cohort-1: organized intervention to patients with DRM or at risk; group 2: intervention on demand by health personnel; Group 3: usual care without any explicit intervention. Effectiveness will be evaluated in relation to multiple outcomes such as: length of hospital stay of the index admission; and the following parameters during admission and until one year after admission, mortality, occurrence of complications (mainly infectious, or surgical in surgical patients), readmissions, use of health resources after discharge (primary care consultations, hospital and emergency consultations), changes in weight during admission and up to one year, changes in their health related quality of life (SF-36 and/or EQ-5d) and fragility (Barthel I.) from admission to one year after admission.
2. -Evaluate the cost and cost-effectiveness of those strategies.
3. - Evaluate in the three groups the evolution of patients in relation to the previous parameters of results according to their classification after screening at the time of admission to DRM, risk of DRM or no problem of DRM detected.

   Secondary Objectives
4. - Evaluate the three groups of patients classified according to their level of DRM according to their level of fragility and in relation to their evolution during admission and up to one year (based on all the outcome parameters indicated above)
5. - Identify risk factors of worse evolution during hospital admission and up to one year of follow up based on the previously described outcome parameters and study the role that the DRM level plays as predictor of evolution.

DESIGN: Prospective cohorts with three branches. SCOPE: Three public hospitals. The first center, where the study intervention will be carried out (branch 1), is the Galdakao - Usánsolo University Hospital that serves a population of about 300,000 urban inhabitants and semi-urban The second center, the University Hospital of Basurto (HUB), where the intervention will be carried out by demand (branch 2), serves the population of Bilbao, some 350,000 urban inhabitants. The third center, Donostia University Hospital (HUD) where there will be no specific organized intervention (branch 3), attends the population of San Sebastián-Donostia and surrounding areas covering a population of about 400,000 inhabitants of urban and semi-urban characteristics. All of them have similar human and technological resources being the population that attend similar on sociodemographic and clinical characteristics.

SUBJECTS OF THE STUDY. See detailed information in other sections. SAMPLE SIZE. It is estimated at least 10-15% of DRM and up to 30-35% of patients at risk of DRM (with a global of almost 40-50%) in the selected pathologies of patients.

Sample size calculation. We have made the estimates for an alpha error of 0.05 and a power of 80%. We have chosen the following outcome parameter in which we expect relevant differences between branches: we estimate that the average length of stay will decrease from an average of 12 days (DS: 5) in the DRM group or at risk without any explicit intervention (HUD) to an average of 10 days (DS: 5) in the DRM group or at risk where the intervention will be performed (HGU) for which we will need 100 patients by each comparisons group but we will try to recruit at least 100 patients from the previous three nutritional groups per center. We estimate a percentage of losses in the follow-up of 10-15% so, overall, 350 patients per center will be sufficient to meet the objectives and respond to the hypotheses of the study. Data from 2017 for each hospital and established patients selection criteria indicate that we should have more than those patients admitted by hospital in 12 months.

DESCRIPTION OF THE SCREENING: all admitted patients of the three centers that meet the selection criteria will be evaluated in the first 72 hours after admission and again upon discharge (if a patient remained admitted more than one week, this assessment will be repeated weekly). The nutritional risk assessment will be done by applying the Malnutrition Universal Screening Tool (MUST) and the Global Leadership Initiative on Malnutrition (GLIM) questionnaires.

VARIABLES TO COLLECT: in summary, A.-From the clinical history: Sociodemographic data will be collected (age, gender, educational level ..) and clinical data such as: comorbidities, based on the Charlson Comorbidity Index , weight, height, health habits, usual treatments (dose, number of drugs), diagnosis of admission (Major Diagnostic Categories ICD-10), severity of pathology (TNM if pathology tumor), source of admission (emergency vs scheduled), admission service. During admission: complications, treatments, procedures and referral to special units (ICU,...). Analytical data available (biochemistry and blood cells count, including urea, creatinine, glucose, electrolytes, albumin, pre-albumin, lymphocytes, total cholesterol, triglycerides, transferrin, and liver function tests). This analytics will be obtained in the first 48 hours of admission and in surgical patients before the intervention if scheduled. They will be repeated at discharge and weekly in prolonged income.

Main results of interest: see separate section. B.-Health-related quality of life questionnaires: 1.- The patient's functional will be calculated using the Barthel index. 2. - General health and utilities: they will be measured by the EuroQol-5d questionnaire, which will mainly be used for economic analysis. 3.-SF-36.

STATISTIC ANALYSIS. A descriptive analysis of the entire sample and univariate analysis to determine potential variables related to the outcomes of interest will be performed. In the multivariable analysis, different models will be used according to the dependent/outcome variable of interest. In the case of dichotomous dependent variables (mortality, complications, readmissions ...) logistic regression models will be used. For continuous dependent variables (changes in HRQoL) generalized linear models will be used; and for dependent variables that have other distributions, such as length of stay, Poisson regression models will be used. The main comparison will be between the intervention groups (HGU) versus intervention by demand (HUB) versus control group (HUD). In all multivariables analyzes, the use of a Propensity Score (PS) as an adjustment system for the differences between the characteristics of the patients of the three centers will be considered.

Economic analysis: A cost-effectiveness analysis of the intervention corresponding to the first branch will be carried out with respect to the second and third branches. Only medical costs associated with medical assistance will be included. The measure for the cost-effectiveness analysis will be the incremental cost for each year of life adjusted by Quality Adjusted Life Year (QALY) earned. The QALY will be calculated from the EuroQol-5d-5l questionnaire scores, in the baseline moment and one year after admission, and the mortality variable up to the year.

PROBLEMS AND LIMITATIONS OF THE STUDY. 1.-As in any study prospective study, main problem is the losses in the follow up. To reduce them, patients will be fully informed and a close contact will be established during follow-up to all patients. 2.-This project is proposed as an intervention study adapted to the current circumstances of the usual clinical care practice, which should guarantee a greater feasibility of a subsequent implementation of this patient care strategy if our results show its benefits. 3.- The comparability between the different cohorts will be guaranteed in the statistical analysis by the adjustment by the propensity scores. 4.-The strategy of the study poses an ethical problem since after screening in all the centers some of the patients will be identified as with DRM or at risk and therefore this will be communicated to the physicians in charge of each patient so that they proceed in the way they create timely by writing down their attitude therapy. We will collect information about any additional nutritional strategy given to any patient.

ETHICAL AND CONFIDENTIALITY ASPECTS. The project has been evaluated and approved by the research commissions of all the participant centers and approved by the accredited Clinical Research Ethics Committee (CEIC) of the Basque Country. EU and Spanish laws on personal data protection will be followed, ensuring that patient information data obtained cannot be associated with identifiable persons. Study data base will be encrypted and protected to assure confidentiality. Only research personal will have access to it with specific passwords.

ELIGIBILITY:
Inclusion Criteria: Patients consecutively admitted to each center in their Digestive, Oncology or Surgery Services and that meet the inclusion criteria and none of the exclusion criteria

* . Pathologies to be included according to ICD 10 criteria : A-Digestive pathologies: acute pancreatitis, ulcerative colitis, Crohn's disease, Inflammatory bowel disease.
* Pathologies to be included according to ICD 10 criteria : .-Oncological pathologies (surgery or admissions at follow up for oncologic patients): esophageal, gastric, colon and rectum cancers , pancreatic cancer, and ulcerative colitis and Crohn's disease admitted with surgical indication.

  -. Patients older than 18 years and who are recruited in the first 48 hours after admission
* . Patients who sign the informed consent.

Exclusion Criteria:

* Patients with serious organic or psychopathological problems or in a terminal situation;
* Patients with neurosensory problems,
* Patients that do not understand the Spanish or Basque language,
* Patients that prevent them from giving their consent
* Patients unable to complete the questionnaires used in the study.
* Patients who are to have surgery by colon or rectum cancers detected by screening (not applicable if they are later admitted by complications of their oncological disease)
* Age under 18,
* Pregnancy,
* Admission to critical units,
* Admission to a short stay unit (<72 hours)
* Admission to a psychiatry,
* Admission to study by weightloss.
* Or those who do not wish to participate or who do not sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1051 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Mean weight changes | Index hospital admission and 12 months follow up
  Mean weight changes from admission to discharge, at hospital at the index admission, and until one year of follow up
Mean length of stay | Index hospital admission
  Mean length of stay at the index admission
Mortality rate | Index hospital admission to 12 months follow up
  Mortality rate at different points in time

SECONDARY OUTCOMES:
Number of Participants with complications | Index hospital admission to 12 months follow up
  Clinical complications, especially infectious complications during admission (CHADx classification) or events during admission, surgical complications (Clavien- Dindo classification ), surgical procedures performed
Number of Participants with Hospital readmissions | Index hospital discharge to 12 months follow up
  Hospital readmissions
Other health care resources use | Index hospital discharge to 12 months follow up
  Number of Participants with primary care consultations, hospital consultations, emergency consultations, separately.
Number of Participants with Adverse effects of the nutrition program | Index hospital admission to12 months follow up
  Infections, Hyperglycemia, Digestive intolerance, Bronchoaspiration, Refeeding syndrome.
Costs | Index hospital admission to12 months follow up
  Monetary costs
Health-related quality of life (HRQoL) changes | Index hospital admission to 12 months follow up
  General HRQoL: It will be measured through the EuroQol-5d questionnaire. Scores from 0 to 100. Higher values indicate best health status
Patient's functional status | Index hospital admission to 12 months follow up
  The patient's functional will be calculated using the Barthel index. Scores 0 to 100. Higher values indicate best functional status

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Covadonga Iglesias, MD, Study Chair — Hospital Universitario Basurto; Alfredo Yoldi, MD, Study Chair — Hospital Donostia
Locations (2):
- Spain (2):
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Galdakao-Usansolo, Galdakao

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be available after main publications
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After december 2024
Access Criteria: By demand and agreement with our institutions

REFERENCES:
- [Background] Bally MR, Blaser Yildirim PZ, Bounoure L, Gloy VL, Mueller B, Briel M, Schuetz P. Nutritional Support and Outcomes in Malnourished Medical Inpatients: A Systematic Review and Meta-analysis. JAMA Intern Med. 2016 Jan;176(1):43-53. doi: 10.1001/jamainternmed.2015.6587. PMID 26720894
- [Background] Cederholm T, Bosaeus I, Barazzoni R, Bauer J, Van Gossum A, Klek S, Muscaritoli M, Nyulasi I, Ockenga J, Schneider SM, de van der Schueren MA, Singer P. Diagnostic criteria for malnutrition - An ESPEN Consensus Statement. Clin Nutr. 2015 Jun;34(3):335-40. doi: 10.1016/j.clnu.2015.03.001. Epub 2015 Mar 9. PMID 25799486
- [Background] Baldwin C, Kimber KL, Gibbs M, Weekes CE. Supportive interventions for enhancing dietary intake in malnourished or nutritionally at-risk adults. Cochrane Database Syst Rev. 2016 Dec 20;12(12):CD009840. doi: 10.1002/14651858.CD009840.pub2. PMID 27996085
- [Background] Parsons EL, Stratton RJ, Cawood AL, Smith TR, Elia M. Oral nutritional supplements in a randomised trial are more effective than dietary advice at improving quality of life in malnourished care home residents. Clin Nutr. 2017 Feb;36(1):134-142. doi: 10.1016/j.clnu.2016.01.002. Epub 2016 Jan 11. PMID 26847947
- [Background] Elia M, Normand C, Norman K, Laviano A. A systematic review of the cost and cost effectiveness of using standard oral nutritional supplements in the hospital setting. Clin Nutr. 2016 Apr;35(2):370-380. doi: 10.1016/j.clnu.2015.05.010. Epub 2015 May 29. PMID 26123475
- [Background] Alvarez-Hernandez J, Planas Vila M, Leon-Sanz M, Garcia de Lorenzo A, Celaya-Perez S, Garcia-Lorda P, Araujo K, Sarto Guerri B; PREDyCES researchers. Prevalence and costs of malnutrition in hospitalized patients; the PREDyCES Study. Nutr Hosp. 2012 Jul-Aug;27(4):1049-59. doi: 10.3305/nh.2012.27.4.5986. PMID 23165541
- [Background] Philipson TJ, Snider JT, Lakdawalla DN, Stryckman B, Goldman DP. Impact of oral nutritional supplementation on hospital outcomes. Am J Manag Care. 2013 Feb;19(2):121-8. PMID 23448109
- [Derived] Martin J, Larrea N, Garcia Y, Bolinaga I, Perales A, Sarasqueta C, Quintana JM. One-year post-discharge health-related quality of life in digestive and oncology patients: a three-group comparison by nutritional status and care. Qual Life Res. 2025 Dec 26;35(1):10. doi: 10.1007/s11136-025-04139-y. PMID 41452524
- [Derived] Garcia Y, Larrea N, Martin J, Bolinaga I, Sarasqueta C, Perales A, Iglesias NC, Yoldi A, Quintana JM; REDISSEC-Malnutrition Research Group. Evaluation of clinical outcomes after an intervention in malnourished hospitalized patients. Clin Nutr. 2025 Nov;54:42-52. doi: 10.1016/j.clnu.2025.04.034. Epub 2025 Sep 18. PMID 41004975